CLINICAL TRIAL: NCT01950169
Title: Effects of Bisphosphonates and Nutritional Supplementation After a Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lena Flodin, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NutristudienSHFG
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2014-09

CONDITIONS: Hip Fracture
Keywords: Hip fracture; Nutritional supplement; Bisphosphonates; Bone mineral density; Body composition
MeSH Terms: conditions — Hip Fractures | interventions — Risedronic Acid; Dietary Supplements; Diphosphonates; Calcium; Cholecalciferol; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Risedronate (Active Comparator): 35 mg risedronate orally administered once weekly for 12 months and orally administered Calcium 1000 mg and 800 IU vitamin D3 daily for 12 months. Group B (bisphosphonate group)
  Interventions: Drug: Risedronate; Dietary Supplement: Calcium and vitamin D3
- Nutritional supplement (Active Comparator): Oral liquid nutritional supplement (600kcal and 40 gram protein/day) for 6 months after the hip fracture besides Risedronate and calcium and vitamin D3. Group BN (bisphosphonate and nutritional supplemented group)
  Interventions: Drug: Risedronate; Other: Nutritional supplement; Dietary Supplement: Calcium and vitamin D3
- Calcium and vitamin D3 (Active Comparator): An oral dose of 1000 mg Calcium and 800 IU vitamin D3 daily for 12 months after hip fracture. Group C (control)
  Interventions: Dietary Supplement: Calcium and vitamin D3

INTERVENTIONS:
Drug: Risedronate — The bisphosphonate group (B) receive 35 mg risedronate (Optinate® Septimum) once weekly for 12 months and calcium (1000 mg) and vitamin D3 (800 IU) (Calcichew-D3®) daily for 12 months.
  Other Names: Bisphosphonate Group (B)
  Arms: Nutritional supplement; Risedronate
Other: Nutritional supplement — The bisphosphonate and nutritional supplemented group (BN) receive 35 mg risedronate once weekly for 12 months plus nutritional supplement (Fresubin® protein energy drink) during the first six months following hip fracture and also calcium (1000 mg) and vitamin D3 (800 IU) daily for 12 months.
  Other Names: Bisphosphonate and nutritional supplemented Group (BN)
  Arms: Nutritional supplement
Dietary Supplement: Calcium and vitamin D3 — The patients in the control group (C) receive orally administered calcium 1000 mg and 800 IU vitamin D3 (Calcichew-D3®) daily for 12 months.
  Other Names: Control Group (C)

SUMMARY:
The study hypothesis is that nutritional supplementation together with bisphosphonates have a better preserving effect on bone mineral density (BMD) after hip fracture than bisphosphonates alone and that nutritional supplementation given postoperatively for 6 months preserve lean body mass in elderly hip fracture patients.

DETAILED DESCRIPTION:
Inclusion criteria: Men and women, ≥ 60 years of age with a recent fracture of the femoral neck or trochanter, admitted to any of the four University hospitals in Stockholm, Sweden. Patients are randomized into three groups by sealed enveloped technique in blocks by 12, thus assuring that each center had an equal distribution of patients in the three treatment groups. Patients randomly assigned and followed for 12 months. Each center with a doctor in charge and a trial nurse. The trial nurse in collaboration with the doctor are responsible of the randomization procedure and that blood samples are taken in the morning of the first weekday after inclusion at the ward and further that the dual-energy X-ray (DXA) and all estimates are done during hospital stay.The pharmacological treatment and nutritional supplementation starts as soon as the patients are circulatory stable, able to take food by mouth and are able to sit in an upright position one hour after taking the tablets.Patients are examined at baseline with a follow up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Recent fracture of the femoral neck or trochanter
* Without severe cognitive impairment
* Ambulant before fracture
* BMI ≤ 28

Exclusion Criteria:

* Abnormal parameters regarding liver i.e. S-Alanine aminotransferase (S-ALAT) and S-Aspartate aminotransferase (S-ASAT) ≥ twice as normal
* Abnormal parameters regarding kidney i.e. S-Creatinine > 130 µg/L
* Primary hyperparathyroidism, osteogenesis imperfecta, Paget´s disease
* Myeloma
* Lactose intolerance
* Dysphagia
* Esophagitis
* Gastric ulcer
* Malignancy
* Diabetes with nephropathy or retinopathy
* Active iritis or uveitis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2004-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Hedström, MD, PhD, Study Director — Karolinska Institutet; Maria Sääf, MD, PhD, Study Director — Karolinska Institutet; Lena Flodin, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Geriatric Medicine R94, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Flodin L, Cederholm T, Saaf M, Samnegard E, Ekstrom W, Al-Ani AN, Hedstrom M. Effects of protein-rich nutritional supplementation and bisphosphonates on body composition, handgrip strength and health-related quality of life after hip fracture: a 12-month randomized controlled study. BMC Geriatr. 2015 Nov 17;15:149. doi: 10.1186/s12877-015-0144-7. PMID 26572609

RESULTS

PARTICIPANT FLOW:
Groups:
- Group B, Bisphosphonates: Patients allocated to intervention B received 35 mg risedronate once weekly for 12 months and 1,000 mg calcium and 800 IU vitamin D3 daily.
- Group BN/N, Bisphosphonates Along With Nutritional Supplementation: Patients allocated to intervention BN/N received 35 mg risedronate once weekly for 12 months plus a nutritional supplement (Fresubin protein energy drink) during the first 6 months after hip fracture. The supplement contained 150 kcal and 10 g protein/100 mL milk-based protein (80 % casein and 20 % whey). Patients were prescribed 200 mL twice daily, totaling 600 kcal with 40 g protein.
- Group C, Control: Patients allocated to group C served as controls and received 1,000 mg Calcium and 800 IU vitamin D3 daily for 12 months.
Period: Overall Study
Arm/Group | Group B, Bisphosphonates | Group BN/N, Bisphosphonates Along With Nutritional Supplementation | Group C, Control
Started | 28 | 26 | 25
Completed | 25 | 18 | 24
Not Completed | 3 | 8 | 1
Not completed — Withdrawal by Subject | 2 | 8 | 1
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group B, Bisphosphonate: Patients were randomized to treatment with bisphosphonates (risedronate 35 mg weekly for 12 months. All patients received calcium (1,000 mg) and vitamin D3 (800 IU) daily.
- C, Control: Patients allocated to group C served as controls and received 1,000 mg Calcium and 800 IU vitamin D3 daily for 12 months.
- Total: Total of all reporting groups
Arm/Group | Group B, Bisphosphonate | Group BN/N, Bisphosphonates Along With Nutritional Supplementation | C, Control | Total
Number analyzed (Participants) | 28 | 26 | 25 | 79
Age, Continuous [Median (Full Range); unit: Years] | 82 [63 to 94] | 82 [62 to 93] | 75 [61 to 96] | 81 [61 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 19 | 56
  Male | 10 | 7 | 6 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Patients who were admitted to one of the four university hospitals in Stockholm, Sweden during 2005-2009, with the diagnosis of femoral neck or trochanteric fracture.
  participants
    Sweden | 28 | 26 | 25 | 79

OUTCOME MEASURES:

1. Primary Outcome: Total Hip Bone Mineral Density (BMD) at Baseline, 6 and 12 Months After Hip Fracture.
Description: Total hip bone mineral density (BMD) was measured by dual-energy X-ray absorptiometry (DXA). The DXA image is two dimensional and BMD was expressed as areal density, grams per square centimeter (g/cm^2). The change in BMD between baseline, 6 and 12 months was registered.
Time Frame: Baseline, 6 months and 12 months
Population: Seventy-nine patients were initially included in the study, of whom 67 were available at final follow-up.
Measure: Mean (Standard Deviation); unit: g/cm^2
Groups:
- B, Bisphosphonate: Patients were randomized to treatment with bisphosphonates (risedronate 35 mg weekly for 12 months. All patients received calcium (1,000 mg) and vitamin D3 (800 IU) daily.
- BN/N, Bisphosphonate Along With Nutritional Supplementation: Patients were randomized to treatment with bisphosphonates along with nutritional supplementation (40 gram protein, 600 kcal daily).
- C, Control: The patients were randomized to receive calcium and vitamin D3 alone and served as controls.
Arm/Group | B, Bisphosphonate | BN/N, Bisphosphonate Along With Nutritional Supplementation | C, Control
Number analyzed (Participants) | 28 | 26 | 25
g/cm^2
  follow up at 6 months: number analyzed (Participants) | 25 | 20 | 25
  follow up at 6 months | -0.008 (0.037) | 0.005 (0.026) | -0.017 (0.026)
  follow up at 12 months: number analyzed (Participants) | 25 | 18 | 24
  follow up at 12 months | -0.012 (0.042) | -0.004 (0.025) | -0.018 (0.032)
Statistical Analysis 1: Comparison: B, Bisphosphonate vs BN/N, Bisphosphonate Along With Nutritional Supplementation vs C, Control; Test type: Superiority; p = 0.05, ANCOVA; Covariates used were age, sex, total mass, and baseline BMD. Data were reported using complete-cases analysis and intention-to-treat (ITT) analysis

2. Primary Outcome: Total Body Mineral Density (BMD) at Baseline, 6 and 12 Months After Hip Fracture.
Description: Total body mineral density (BMD) were assessed by dual-energy X-ray absorptiometry (DXA). The DXA image is two dimensional and BMD was expressed as areal density, grams per square centimeter (g/cm^2). The change in BMD between baseline, 6 and 12 months was registered.
Time Frame: Baseline, 6 months and 12 months
Population: Seventy-nine patients were initially included in the study, of whom 67 were available at final follow-up.
Measure: Mean (Standard Deviation); unit: g/cm^2
Groups:
- B, Bisphosphonate: Patients were randomized to treatment with bisphosphonates (risedronate 35 mg weekly for 12 months. All patients received calcium (1,000 mg) and vitamin D3 (800 IU) daily. Total hip and total body BMD were assessed with dual-energy X-ray absorptiometry at baseline, 6.and 12 months.
Arm/Group | B, Bisphosphonate | BN/N, Bisphosphonate Along With Nutritional Supplementation | C, Control
Number analyzed (Participants) | 28 | 26 | 25
g/cm^2
  follow-up at 6 months: number analyzed (Participants) | 25 | 20 | 25
  follow-up at 6 months | -0.005 (0.018) | -0.006 (0.018) | -0.012 (0.019)
  follow-up at 12 months: number analyzed (Participants) | 25 | 18 | 24
  follow-up at 12 months | -0.003 (0.022) | 0.0006 (0.019) | -0.017 (0.020)
Statistical Analysis 1: Comparison: B, Bisphosphonate vs BN/N, Bisphosphonate Along With Nutritional Supplementation vs C, Control; Test type: Superiority; p = 0.05, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Body Composition, Including Lean Mass at Baseline, 6 and 12 Months After Hip Fracture.
Description: Total body composition, including lean mass composed of muscle, visceral organs and water (LM), fat mass (FM) and bone mineral content (BMC) was measured by dual-energy X-ray absorptiometry (DXA) at baseline and at 6 and 12 months follow up. The sum of lean mass (LM) and BMC represents fat-free mass (FFM). To normalize for body size, FFM was divided by height squared to calculate fat-free mass index (FFMI, kg/m^2).
Time Frame: Baseline, 6 and 12 months
Population: Seventy-nine patients were initially included in the study, of whom 67 were available at final follow-up. Calculations revealed that a sample size of 40 patients per group was required to detect a difference in lean mass between groups (power = 80 %, a = 0.05). However, the study was closed after 4 years due to difficulties in recruiting patients and the study was switched to an exploratory design.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | B, Bisphosphonate | BN/N, Bisphosphonate Along With Nutritional Supplementation | C, Control
Number analyzed (Participants) | 28 | 26 | 25
kg/m^2
  follow up at 6 months | -0.4 (1.2) | -0.9 (0.7) | -0.4 (0.8)
  follow up at 12 months | -0.5 (1.2) | -0.8 (0.9) | -0.5 (0.8)
Statistical Analysis 1: Comparison: B, Bisphosphonate vs BN/N, Bisphosphonate Along With Nutritional Supplementation vs C, Control; Test type: Superiority; p = 0.05, ANCOVA; The analyses included exposure measures treatment groups and sex as fixed factors. Age and baseline values for FFMI, FMI were included as covariates

4. Secondary Outcome: Body Composition, Including Fat Mass at Baseline, 6 and 12 Months After Hip Fracture.
Description: Total body composition, including lean mass composed of muscle, visceral organs and water (LM), fat mass (FM) and bone mineral content (BMC) was measured by dual-energy X-ray absorptiometry (DXA) at baseline and at 6 and 12 months follow up.To normalize for body size, FM was divided by height squared to calculate fat mass index (FMI, kg/m^2).
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | B, Bisphosphonate | BN/N, Bisphosphonate Along With Nutritional Supplementation | C, Control
Number analyzed (Participants) | 28 | 26 | 25
kg/m^2
  follow up at 6 months | -0.6 (1.4) | 0.1 (0.8) | -0.1 (0.8)
  follow up at 12 months | -0.3 (1.6) | 0.1 (0.8) | -0.1 (1.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected 1 year for every patient included.
Description: Once a month the study research nurse interviewed patients by telephone regarding compliance, general state of health and collected adverse event information.
Arm/Group | B, Bisphosphonate | BN/N, Bisphosphonate Along With Nutritional Supplementation | C, Control
All-Cause Mortality (participants affected / at risk) | 1/28 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 2/28 | 0/26 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B, Bisphosphonate (N=28) | BN/N, Bisphosphonate Along With Nutritional Supplementation (N=26) | C, Control (N=25)
Constipation/diarrhea (Gastrointestinal disorders) | 2 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No